CLINICAL TRIAL: NCT03965312
Title: Pilot Clinical Assessment of Low-cost Infant Incubator in Monitoring Temperature and Treating Hypothermia in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: William Marsh Rice University (Other)
Collaborators: Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IncuBaby-NHSRC
Record Dates: First submitted 2019-01-31; First posted 2019-05-29 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Neonatal Hypothermia
MeSH Terms: interventions — Monitoring, Physiologic

STUDY DESIGN:
Intervention Model Description: In the first phase of the study, a novel neonatal temperature monitor and a commercially available patient monitor (Philips Intellivue MP30) will be applied to the same infant; results between them will be compared.
  In the second phase of the study, infants at risk for hypothermia will be placed in an infant incubator; the accuracy of the temperature sensor, time required for infant to become normothermic, and the proportion of time that the infant remains normothermic will be measured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temperature monitoring (1) and incubator test (2) groups (Experimental): In the first (1) phase of the study, the temperature probe and monitor will be attached to infants along with the Philips Intellivue patient monitor. Temperature will be monitored continuously for up to 72 hours.
  In the second (2) phase of this study, infants at risk for hypothermia and not eligible for skin-to-skin care will be placed in the incubator.
  Interventions: Device: Continuous temperature monitor; Device: Neonatal Incubator; Device: Patient monitor

INTERVENTIONS:
Device: Continuous temperature monitor — Temperature will be measured using a novel temperature monitor continuously for up to 72 hours. Accuracy (as compared to a commercially available patient monitor) will be evaluated.
  Other Names: IncuBaby temperature sensor and monitor; Neonatal temperature monitor
Device: Neonatal Incubator — Infants at risk for hypothermia will be placed in a neonatal incubator. Their temperature will be monitored as they are treated. The infant will be treated until the infant is transitioned to skin-to-skin care, discharged, or no longer at risk for hypothermia.
  Other Names: IncuBaby
Device: Patient monitor — Temperature will be measured using a commercially available patient monitor.
  Other Names: Philips Intellivue patient monitor

SUMMARY:
A team of researchers at Rice University and Queen Elizabeth Central Hospital (QECH) are working to develop a low-cost infant incubator called "IncuBaby" that consists of two components: a temperature sensor that can continuously monitor an infant's temperature, and a heated, enclosed area that can adjust internal temperature based on the feedback from the temperature sensor. This robust, low-cost device will allow for the individualized treatment of hypothermia with minimal intervention from the clinical staff. In this study, researchers intend to evaluate the efficacy of this incubator at QECH by comparing infants' temperatures before and after treatment, and calculating the proportion of time that the infants remain in a normothermic range after rewarming. During phase I of this study, the infants will be continuously monitored using the IncuBaby temperature sensor and a gold standard temperature monitor for up to 3 days. The accuracy of the IncuBaby temperature sensor will be determined by calculating the difference between the temperatures recorded by the temperature sensor and the commercial patient monitor at each point in time. During phase II of the study, infants in need of thermal care with an incubator will be treated with an IncuBaby device and their temperatures will be continuously monitored by both the temperature sensor of the IncuBaby device and a commercially available patient monitor. Care will continue at the clinician's discretion until the infant can be weaned from the incubator or until patients are withdrawn from the study and placed on the standard of care. To determine the effectiveness of the IncuBaby device at warming infants, the temperatures of the infants will be compared before and after treatment for each subject. The proportion of time the device maintains the subject's temperature in a normal range will also be calculated.

DETAILED DESCRIPTION:
This is a two-phase, pilot prospective study to determine the effectiveness of a low-cost incubator in warming infants and regulating their temperatures. The temperature sensor that controls the heat of the incubator based on the infant's temperature has been previously evaluated in Rice IRB approved studies in Houston, TX with plans to evaluate at QECH. The first phase will validate the use of the temperature sensor in infants by comparing it to a commercial temperature monitor. The second phase will test the effectiveness of the IncuBaby device using that temperature sensor to regulate the heat of the infant.

Treatment and Monitoring of Neonates

During Phase I, the following steps will be taken:

A trained study nurse will assess the subject for clinical complications before attaching the temperature monitoring device.

A trained study nurse or clinician will attach the temperature monitoring device to the infant. A trained research assistant from Rice University or from the Biomedical Engineering Department at Malawi Polytechnic will observe all procedures and will notify the nurse of any observed errors so they may be corrected. They will also be able to answer any technical questions from the nurse.

The trained study nurse will attach the temperature probe from the commercial patient monitor as well as provide any other care needed.

A research assistant will use a laptop to collect the electrical signals from both temperature monitors.

Temperature monitoring will continue for up to 3 days. The research assistant may ask the nurse to remove and reapply the temperature monitor during this period.

Upon removal of the abdominal strap at the end of the study, the subject may be monitored for up to one hour in order to assess the effect of the abdominal strap on the skin of the subject.

Once Phase I is complete, Phase II will begin. During Phase II, the following steps will be taken:

A trained study nurse will assess the subject for clinical complications before beginning treatment.

A trained study nurse or research technician will turn the incubator on to begin pre-warming.

A trained study nurse or clinician will attach the temperature probe from the IncuBaby device to the infant and then place the infant in the incubator. A trained research assistant from Rice University or from the Biomedical Engineering Department at Malawi Polytechnic will observe all procedures and will notify the nurse of any observed errors so they may be corrected. They will also be able to answer any technical questions from the nurse.

The trained study nurse will attach the temperature probe from the commercial patient monitor as well as provide any other care needed.

A research assistant will use a laptop to collect the data from both devices.

Care will be continued at the discretion of the clinician until the infant can be weaned from the IncuBaby device. The infant may be weaned to the standard of care or end thermal treatment. The infant will be transitioned to KMC as soon as possible after these eligibility criteria are fulfilled:

Completed other treatment (CPAP, phototherpay, IV) Mom/caregiver becomes available Weight increases > 1000 g Becomes clinically stable Body temperture is stable and not dipping below normal despite thermal support

Based on the discretion of the clinician, the subject may be weaned to KMC or an open cot. The IncuBaby device has a "weaning" setting that turns off the heaters in the incubator but continues to monitor the infant's temperature. If the infant is found to be hypothermic after ending treatment and the clinician recommends continued incubator care, the subject may recommence use of the IncuBaby for treatment.

The commercial patient monitor will alert nursing staff if the baby's temperature becomes too high or too low. Temperature settings for alarms will be set by a clinician so that the high temperature alarm is > 37.5 C, and the low temperature alarm is < 36.5 C. During Phase II, the following steps will be recommended if the commercial patient monitor sounds a high or low temperature alarm. These guidelines were written in accordance with current clinical practice at QECH. The study nurse can also choose to discontinue the use of the IncuBaby device at any time.

High temperature alarm - indicates possible hyperthermia Check that the incubator temperature is at 36C or less. Open the incubator and recheck the baby's temperature If baby's temperature is still above normal remove blankets/clothing If baby is febrile despite these measures look for a clinical reason for the temperature Remove the infant from the IncuBaby device Low temperature alarm - indicates possible hypothermia

Check that the incubator is in on and functioning Check that the temperature probe has not fallen off. Recheck the baby's temperature If temperature still low add blankets/clothing and hat If the temperature is still low look for a clinical reason for the hypothermia

During both phases, a research assistant will be available during the trial to mitigate any complications with the device. A nurse will be available to respond to alarms from the continuous patient monitor. If the subject's guardian, the nurse, or the research assistant indicates concern during the tests, the study treatment can be discontinued and the subject will return to the standard of care.

Intended Data Collection:

Clinical data will be collected on paper forms as is consistent with current clinical practice. Data will be saved on a secure study server for analysis. Clinical and/or research personnel will record information, excluding personal identifiers, on a standardized patient monitoring form. After the subject's participation is complete, a research assistant will collect and scan the form. We will collect the following information:

1. Baseline demographic and relevant medical information

   a. Recorded one at enrollment i. Date of study ii. Date of birth iii. Sex iv. Birth weight v. Type of delivery vi. Gestational age at birth vii. Corrected gestational age viii. Abdominal circumference ix. Admission temperature b. Recorded throughout study as clinically collected i. Other comorbidities ii. Medications/treatments given iii. Current weight iv. Temperature measurements taken as standard of care
2. Accuracy a. Recorded automatically by study equipment i. Abdominal temperature from IncuBaby temperature probe and gold standard device ii. Alarms iii. Temperature in incubator* b. CO2 levels c. Humidity levels in the incubator d. Movement/other caregiving e. Fit/tightness of the strap during and/or at end of study f. Ambient temperature g. Routine assessment of abdominal skin (i.e. indentation, skin irritation) h. Strap site assessment during and/or at end of study i. Commercially available patient monitor temperature sensor site assessment during and/or at end of study j. Nurse comments k. Research technicians comments

   * Phase II only, if enclosed A log of an observed user error or comments about the device will be used to improve future iterations of the device. The nurse and technician monitoring forms that will be used to record the above variables are attached to this proposal.

ELIGIBILITY:
Inclusion Criteria:

* The subject is currently being treated at QECH in the neonatal ward.
* An IncuBaby device and study monitor are available for use.
* The subject's caregiver has provided informed consent for their child to participate (consent form attached to this proposal).
* Phase II only: the subject is eligible for thermal care in an incubator. If the subject is recommended for KMC, they will not be eligible for participation in this study. To be considered for care with the IncuBaby, infants should be:

  * Less than 1000 g
  * Or > 1000 g but

    * Receiving medical interventions such as CPAP, oxygen, phototherapy, or IV
    * Unstable, critically ill or surgical conditions
    * No mother or caregiver available for KMC
    * Mother too sick to provide KMC
    * Clinician in charge has decided against KMC as requires closer supervision by nursing staff
    * No space in KMC

Exclusion Criteria:

The subject may be excluded from the study at the clinician's discretion for any reason including potential for skin irritation, cough or other condition that may preclude use of the temperature belt, or concurrent treatments that may require increased patient care. Only subjects eligible for care in an incubator will be enrolled in phase II.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2017-07-31 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Temperature monitor accuracy | from time of enrollment until intervention is complete; up to 28 days
  Continuously measured temperature for temperature monitor compared against Philips Intellivue patient monitor
Temperature of incubator | from time of enrollment until intervention is complete; up to 28 days
  Continuously measured temperature of incubator
Temperature of infant | from time of enrollment until intervention is complete; up to 28 days
  Continuously measured temperature of infant

SECONDARY OUTCOMES:
Time until normothermia | from time of enrollment until intervention is complete; up to 28 days
  Time until infant becomes normothermic (36.5-37.5C)
Proportion of time normothermic | from time of enrollment until intervention is complete; up to 28 days
  The proportion of treatment time that the infant is normothermic (36.5-37.5C)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Richards-Kortum, PhD, Principal Investigator — William Marsh Rice University; Queen Dube, MD, Principal Investigator — Kamuzu University of Health Sciences
Locations (1):
- Queen Elizabeth Central Hospital, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sosa Saenz SE, Hardy MK, Heenan M, Oden ZM, Richards-Kortum R, Dube Q, Kawaza K. Evaluation of a continuous neonatal temperature monitor for low-resource settings: a device feasibility pilot study. BMJ Paediatr Open. 2020 May 7;4(1):e000655. doi: 10.1136/bmjpo-2020-000655. eCollection 2020. PMID 32426530

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT03965312/Prot_SAP_001.pdf
  • Informed Consent Form (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT03965312/ICF_000.pdf